CLINICAL TRIAL: NCT01961583
Title: Evaluation of [18F]FluciclatidePositron Emission Tomography For the Prediction of Response to Pazopanib In Patients With Metastatic Renal Cell Carcinoma: An Exploratory Study
Brief Title: [18F]Fluciclatide PET Imaging of Pazopanib Response
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination of [18F]Fluciclatide production
Sponsor: Asan Medical Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Jin-Sook Ryu, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-0382
Record Dates: First submitted 2013-10-07; First posted 2013-10-11 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Kidney Neoplasm
MeSH Terms: conditions — Kidney Neoplasms | interventions — AH 111585

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug; 18F-Fluciclatide (Experimental): 18F-Fluciclatide, 0.14 mCi/kg (not to exceed 10 mCi), IV(in the vein) administration
  Interventions: Drug: 18F-Fluciclatide

INTERVENTIONS:
Drug: 18F-Fluciclatide — Baseline 18F-Fluciclatide PET imaging will be obtained before starting of Pazopanib therapy(within 7 days).
  Subsequent 18F-Fluciclatide PET should be performed on 7 days after Pazopanib therapy
  Other Names: AH111585

SUMMARY:
Positron emission tomography (PET) is a non-invasive imaging tool for monitoring functional and metabolic responses of biological events with specific radiotracer in vivo. The PET tracer [18F]Fluciclatide is an 18F radiolabeled small peptide containing the RGD (arginine-glycine-aspartate) tri-peptide, which preferentially binds with high affinity to αvβ3 and αvβ5 integrins. αvβ3-integrins are expressed at low levels on epithelial cells and mature endothelial cells but are expressed at high levels on activated endothelial cells in the neo-vasculature of a range of tumors and it also may regulate angiogenesis. If pazopanib acts mainly on active angiogenetic tumors, the quantitative uptake of [18F]Fluciclatide can be used to predict the effect of this antiangiogenic drug. The investigators expected the baseline tumor uptake in [18F]Fluciclatide to be able to predict treatment response, and planned a study of [18F]FluciclatidePET for patients with metastatic RCC who received pazopanib systemic therapy.

DETAILED DESCRIPTION:
Subjects will receive treatment with pazopanib at a dose of 800 mg orally once daily. [18F]Fluciclatide imagings will be taken 2 times; 1) before systemic therapy (at baseline), 2) at one week after starting of Pazopanib. However, If the target lesion on the baseline PET cannot be discriminated compared to the background activity, the 2nd PET will not be done. Response evaluation by CT will be performed at baseline, at 6 week, at 12 week and every 8 weeks thereafter until the end of treatment. RECIST1.1 criteria for response will be applied. Patient will be treated with Pazopanib until there is disease progression, unacceptable toxicity or withdrawal of patient consent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed renal cell carcinoma, stage IV patient.
* The tumor mass ≥1.5cm in diameter that is planned to receive Pazopanib as systemic antiangiogenic therapy.
* Pretreatment CT with or without contrast within 4 weeks prior to the first 18F-Fluciclatide PET scan.
* Evidence of unidimensionally measurable lesion(s) by RECIST criteria version 1.1.
* No prior systemic anti-angiogenic therapy for metastatic disease; prior antiangiogenic therapy used as an adjuvant therapy is allowed if it is completed 6 or more months before study enrollment.
* Male or female aged over 20 years
* Be ambulatory and have an Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Have a life expectancy of at least 3 months.
* Adequate medical condition in the judgment of the investigator
* Be willing and able to comply with the protocol for the duration of the study.
* Be willing and able to implement effective contraceptive practice
* Give written informed consent prior to study-specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

* Received another IMP within 30 days before the first administration of 18F-Fluciclatide injection.
* Inability to perform 18F-Fluciclatide PET imaging studies due to physical inability or claustrophobia.
* Intra-hepatic tumor only (without extra-hepatic tumor)
* Chemotherapy within 2weeks, or received radiotherapy to the region of the target lesion, surgery of target lesion within 2 weeks prior to the first 18F-Fluciclatide PET scan
* Pregnant, nursing women or patients with reproductive potential without contraception.
* Current treatment on another therapeutic clinical trial(except Pazopanib study)
* Any patients with known allergy to the GE health care product or any or its excipients should be excluded from the study
* Any condition that, in the opinion of the investigator, would compromise the well-being of the subject or the study or prevent the subject from meeting or performing study requirements.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Baseline 18F-Fluciclatide PET SUV | Prior to starting Pazopanib treatment
  The difference of the baseline 18F-Fluciclatide PET SUV between responders and non-responders by RECIST criteria after Pazopanib therapy

SECONDARY OUTCOMES:
The difference of 18F-Fluciclatide PET parameters (% change of SUV) between responders and non-responders by RECIST criteria | 7±1 days after Pazopanib treatment
Progression free survival more than 6 month | More than 6 month after 1st PET scan
  Progression free survival defined as time from PET scan to the date of death, recurrence or progression

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Sook Ryu, MD. PhD., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, Songpa-gu, South Korea

REFERENCES:
- See also: Cancer, Nuclear Scans — http://www.nlm.nih.gov/medlineplus
- See also: Pazopanib — http://druginfo.nlm.nih.gov/drugportal/drugportal.jsp